CLINICAL TRIAL: NCT02264977
Title: Evaluation of the GORE® TAG® Thoracic Branch Endoprosthesis (Branched TAG® Device) in the Treatment of Aortic Arch Aneurysms
Brief Title: Early Feasibility of the Branched TAG® Device in the Treatment of Aortic Arch Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SSB 11-03
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Aneurysm of Aortic Arch
MeSH Terms: conditions — Aneurysm, Aortic Arch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Branched TAG® Device (Experimental): Treatment with the GORE® TAG® Thoracic Branch Endoprosthesis
  Interventions: Device: GORE® TAG® Thoracic Branch Endoprosthesis

INTERVENTIONS:
Device: GORE® TAG® Thoracic Branch Endoprosthesis

SUMMARY:
The purpose of this study is to assess the early feasibility of the use of the GORE® TAG® Thoracic Branch Endoprosthesis to treat aneurysms involving the aortic arch

DETAILED DESCRIPTION:
The GORE® TAG® Thoracic Endoprosthesis (TAG® Device) received premarket approval (PMA) for use in endovascular aneurysm repair of the descending thoracic aorta (DTA) on 23-Mar-2005 under P040043, and design changes that resulted in the conformable GORE® TAG® Thoracic Endoprosthesis (CTAG) received premarket approval for the treatment of aneurysms of the DTA on 23-Aug-2011 (P040043/S039). The TAG® Device and CTAG are intended to exclude an aneurysm from the blood circulation in patients diagnosed with DTA aneurysms. However, endovascular treatment options for patients with aortic arch aneurysms are limited as current stent graft technology would require coverage of aortic arch vessels. This prompted the creation of the GORE® TAG® Thoracic Branch Endoprosthesis (previously known as Branched TAG® Device), which was being evaluated under IDE G130120 for Zone 2 aneurysms when this clinical investigation was initiated to evaluate the GORE® TAG® Thoracic Branch Endoprosthesis for the treatment of Zone 0 and Zone 1 aneurysms of the aortic arch.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of aortic aneurysm involving the aortic arch deemed to warrant surgical repair which requires proximal graft placement in Zone 0 or Zone 1:

   1. Fusiform (≥ 55 mm), or
   2. Fusiform (>2 times native aortic diameter), or
   3. Saccular (no diameter criteria)
2. Subject is considered a high risk candidate for conventional open surgical repair at the discretion of the Investigator
3. Age ≥18 years at time of informed consent signature
4. Subject is capable of complying with protocol requirements, including follow-up
5. Informed Consent Form (ICF) is signed by Subject or legal representative
6. Must have appropriate proximal aortic landing zone, defined as:

   1. Must require placement of the proximal extent of the Aortic Component in Zone 0 or Zone 1 for exclusion of the lesion
   2. Acceptable proximal landing zone outer curvature length for the required device
   3. Landing zone inner diameters between 16-48 mm in Zone 1 Subjects and 24-48mm in Zone 0 Subjects
   4. Landing zone, which must include either the brachiocephalic or left common carotid native ostium, cannot be aneurysmal, heavily calcified, or heavily thrombosed
7. Must have appropriate distal aortic landing zone, defined as:

   1. Outer curvature length must be ≥2cm proximal to the celiac artery
   2. Aortic inner diameters between 16-48 mm (diameter must be between 16-42mm if using distal TAG® Device extension)
   3. Landing zone cannot be aneurysmal, heavily calcified, or heavily thrombosed
   4. Landing zone in native aorta or previously implanted GORE® TAG® Device
8. Must have appropriate target branch vessel landing zone, defined as:

   1. Length of ≥3 cm proximal to first major branch vessel if using Aortic Component with 8 mm portal diameter, or length of ≥2.5 cm proximal to first major branch vessel if using Aortic Component with 12 mm portal diameter (required for Zone 0 Subjects)
   2. Target branch vessel inner diameters of 6-15 mm if using Aortic Component with 8mm portal diameter, or inner diameters of 11-18 mm if using Aortic Component with 12mm portal diameter (required for Zone 0 Subjects)
   3. Target branch vessel landing zone must be in native aorta that cannot be aneurysmal, heavily calcified, or heavily thrombosed

Exclusion Criteria:

1. Concomitant aneurysm/disease of the ascending aorta, or abdominal aorta requiring repair
2. Previous endovascular repair of the ascending aorta
3. Previous endovascular repair of the DTA with a non-Gore device
4. Surgery within 30 days of treatment
5. Infected aorta
6. Dissection of the aorta
7. Intramural hematoma of the aortic arch or DTA without aneurysm
8. Life expectancy <2 years
9. Myocardial infarction or stroke within 6 weeks prior to treatment
10. Patient has a systemic infection and may be at increased risk of endovascular graft infection
11. Pregnant female at time of informed consent signature
12. Degenerative connective tissue disease, e.g. Marfan's or Ehler-Danlos Syndrome
13. Participation in another drug or medical device study within one year of study enrollment
14. Known history of drug abuse within one year of treatment
15. Significant thrombus or atheroma in the aortic arch
16. Tortuous or stenotic iliac and/or femoral arteries preventing introducer sheath insertion and the inability to use a conduit for vascular access
17. Planned coverage of celiac artery
18. Patient has known sensitivities or allergies to the device materials
19. Patient has known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment
20. Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin
21. Diameter taper outside of the device sizing range between proximal and distal landing zones of aorta and the inability to use additional devices of different diameters to compensate for the taper
22. Mycotic aneurysm
23. Persistent refractory shock (systolic blood pressure <90 mm Hg)
24. Patient has body habitus or other medical condition which prevents adequate visualization of the aorta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2022-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Dake, MD, Principal Investigator — Stanford University
Locations (6):
- United States (6):
  - Leland Stanford Junior University, Stanford, California
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The Hitchcock Foundation (Dartmouth Hitchcock Medical Center), Lebanon, New Hampshire
  - Hospital at University of Pennsylvania, Philadelphia, Pennsylvania
  - Univerisity of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Branched TAG® Device: Treatment with the GORE® TAG® Thoracic Branch Endoprosthesis
  Branched TAG® Device
Period: Overall Study
Arm/Group | Branched TAG® Device
Started | 9
Completed | 4
Not Completed | 5
Not completed — Death | 3
Not completed — Physician Decision | 1
Not completed — Refuse to return | 1

BASELINE CHARACTERISTICS:
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
BMI, Continuous [Mean (Standard Deviation); unit: kg/(m^2)] | 26.2 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Study Device Access
Description: Access to the aneurysm and target landing zone location is obtained via conventional vascular access and endovascular techniques.
Time Frame: During treatment procedure (day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: Number of Participants With Successful Study Device Deployment
Description: Absence of deployment failure will be considered a successful deployment. Deployment failure will be considered the failure of any Branched TAG® Device component (Aortic Component, Aortic Extender, or SB Component) to be released from the delivery catheter resulting in a serious adverse event (SAE) due to mechanical failure or use error.
Time Frame: During treatment procedure (day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 9
Participants | 9

3. Primary Outcome: Number of Participants With Primary Procedural Side Branch Patency
Description: The presence of forward flow through the implanted Side Branch Component into the target branch vessel.
Time Frame: At conclusion of the treatment procedure (day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 9
Participants | 9

4. Secondary Outcome: Number of Participants With 1 Month Side Branch Primary Patency Assessed by an Independent Core Lab
Time Frame: 1 Month
Population: One participant not assessed for patency at 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 8
Participants | 8

5. Secondary Outcome: Number of Participants Without 1 Month Device Related Endoleaks Assessed by an Independent Core Lab
Description: Device-related endoleaks are defined as the presence of contrast within the aneurysm sac originating from the junction between any Branched TAG® Device component and the landing zone (Type IA or IB) or the junction between the Aortic Component and either the Side Branch Component or the Aortic Extender (Type III).
Time Frame: 1 Month
Population: Two participants not assessed for endoleaks at 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: From endovascular procedure through 60 months
Arm/Group | Branched TAG® Device
All-Cause Mortality (participants affected / at risk) | 3/9
Serious Adverse Events (participants affected / at risk) | 9/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Branched TAG® Device (N=9)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Congestive cardiac failure aggravated (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
Systolic heart failure (Cardiac disorders) | 1 (1)
Hemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Physical deconditioning (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Diverticulitis of colon with hemorrhage (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Mediastinal infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Staphylococcal bacteremia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Lumbar vertebral fracture L2 (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Pseudogout (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 1 (1)
Arm spasticity (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular infarction (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Middle cerebral artery stroke (Nervous system disorders) | 1 (1)
Numbness of lower extremities (Nervous system disorders) | 1 (1)
Numbness of upper arm (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis leg (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Branched TAG® Device (N=9)
Acute post hemorrhagic anemia (Blood and lymphatic system disorders) | 2 (2)
AV block first degree (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 2 (3)
Left atrial appendage thrombosis (Cardiac disorders) | 1 (1)
Mobitz type I (Cardiac disorders) | 1 (1)
Right bundle branch block (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Transient visual loss (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (non-cardiac) (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fever of unknown origin (General disorders) | 1 (1)
Neck swelling (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Stent-graft endoleak type II (General disorders) | 2 (2)
Acute cystitis (Infections and infestations) | 1 (1)
Candidemia (Infections and infestations) | 1 (1)
Cellulitis of leg (Infections and infestations) | 1 (1)
Lower urinary tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ankle sprain (Injury, poisoning and procedural complications) | 1 (1)
Bruise of head (Injury, poisoning and procedural complications) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1)
Contusion of chest wall (Injury, poisoning and procedural complications) | 1 (1)
Contusion of elbow (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fractured toe (Injury, poisoning and procedural complications) | 1 (1)
Laceration of face (Injury, poisoning and procedural complications) | 1 (1)
Laceration of wrist (Injury, poisoning and procedural complications) | 1 (1)
Neck sprain (Injury, poisoning and procedural complications) | 1 (1)
Rib contusion (Injury, poisoning and procedural complications) | 1 (2)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Gout acute (Metabolism and nutrition disorders) | 1 (1)
Calf pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign esophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Apraxia (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Dizziness exertional (Nervous system disorders) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 1 (1)
Foot drop (Nervous system disorders) | 1 (1)
Hemiparesis (right) (Nervous system disorders) | 1 (1)
Incoordination (Nervous system disorders) | 1 (1)
Numbness in leg (Nervous system disorders) | 1 (1)
Paralysis arm (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Weakness left or right side (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Anxiety depression (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No